CLINICAL TRIAL: NCT00506727
Title: A Randomized, Double-Blind, Parallel-Group, Analog Classroom Study, Evaluating ADDERALL XR Versus STRATTERA, Dosed Once Daily, in Children Aged 6-12 With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Analog Classroom Study Comparison of ADDERALL XR With STRATTERA in Children Aged 6-12 With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLI381-404
Record Dates: First submitted 2007-07-19; First posted 2007-07-25 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — SLI381; Atomoxetine Hydrochloride

ARMS (2):
- Adderall XR (Experimental)
  Interventions: Drug: Mixed amphetamine salts (ADDERALL XR)
- Atomoxetine hydrochloride (Active Comparator)
  Interventions: Drug: Atomoxetine hydrochloride

INTERVENTIONS:
Drug: Mixed amphetamine salts (ADDERALL XR)
  Arms: Adderall XR
Drug: Atomoxetine hydrochloride
  Other Names: Strattera
  Arms: Atomoxetine hydrochloride

SUMMARY:
Evaluate the behavioral effects of ADDERALL XR versus STRATTERA under controlled conditions utilizing the SKAMP deportment scale.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of ADHD combined subtype or predominantly hyperactive-impulsive subtype, based on psychiatric evaluation
* Capable of understanding and following classroom instructions
* Generally functioning academically at age-appropriate levels

Exclusion Criteria:

* ADHD, predominantly inattentive subtype
* Controlled or uncontrolled comorbid psychiatric diagnosis (except ODD) with significant symptoms such as PTSD, psychosis, bipolar disease, severe OCD, severe depressive or severe anxiety disorder
* Documented history of aggressive behavior serious enough to preclude participation in regular classroom activities
* Documented allergies or intolerance to either of the active treatments or tricyclic antidepressants

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2003-08-05 (Actual); Primary Completion 2004-07-02 (Actual); Study Completion 2004-07-02 (Actual)

PRIMARY OUTCOMES:
Change in SKAMP deportment scores from baseline to endpoint (averaged across Days 7, 14, 21) | Approximately 3 weeks

SECONDARY OUTCOMES:
PERMP, SKAMP attention scale, CGI, CGIS-P, Peds QL | Approximately 3 weeks
treatment-emergent adverse events | approximately 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Wigal SB, McGough JJ, McCracken JT, Biederman J, Spencer TJ, Posner KL, Wigal TL, Kollins SH, Clark TM, Mays DA, Zhang Y, Tulloch SJ. A laboratory school comparison of mixed amphetamine salts extended release (Adderall XR) and atomoxetine (Strattera) in school-aged children with attention deficit/hyperactivity disorder. J Atten Disord. 2005 Aug;9(1):275-89. doi: 10.1177/1087054705281121. PMID 16371674
- See also: FDA-approved labelling information, US only — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.Label_ApprovalHistory
- See also: FDA Recall information — http://www.fda.gov/opacom/7alerts.html